CLINICAL TRIAL: NCT05368766
Title: Predictive Value of Venous Excess Ultrasound Score in Management of Cardiorenal Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Ayad Habib Said, Principal Investigator, Assiut University
Other Study IDs: VExUS score in cardiorenal
Record Dates: First submitted 2022-04-13; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Cardio-Renal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Diuretics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VExUS score — The venous excess ultrasound (VExUS) score incorporates hepatic venous, intrarenal venous Doppler, inferior vena cava (IVC) assessment, and portal vein Doppler
Drug: Diuretic Effect — Response to diuretic therapy

SUMMARY:
To assess predictive value of venous excess ultrasound score in cardiorenal patient management

DETAILED DESCRIPTION:
Cardiorenal syndrome encompasses a spectrum of disorders involving both the heart and kidneys in which acute or chronic dysfunction in 1 organ may induce acute or chronic dysfunction in the other organ.

Fluid overload is deleterious in critically ill patients; apart from increased mortality, it can cause end-organ damage, thereby increasing the incidence of acute kidney injury (AKI), length of stay in ICU, and duration of mechanical ventilation.

Elevation of central venous pressure is directly transmitted to the renal veins because venous vascular resistance is negligible. As the encapsulated kidney has little room to expand, venous congestion causes renal interstitial hydrostatic pressure to increase. Furthermore, as the post-glomerular vascular and tubular network is a low-pressure system , the increase in the renal interstitial pressure causes compression or even occlusion of renal tubules. That in turn results in reduction or even shut down of tubular flow and shut down in the glomerular filtration .

The venous excess ultrasound (VExUS) score incorporates hepatic venous, intrarenal venous Doppler, inferior vena cava (IVC) assessment, and portal vein Doppler. By utilizing multiple parameters, the negative aspects of individual parameters might get negated and could be considered as a reliable tool to assess congestion of kidneys.

The investigators hypothesise that VExUS score could be valuable in predicting cardiorenal patients who need ultrafiltration in ICU. In this study the investigators will use VEXSUS score to predict response to diuretic therapy, to evaluate patients' volume status, and to predict mortality in cardiorenal patient

Every patient will be subjected to

1. Medical history taking.
2. Complete physical examination.
3. Routine laboratory investigations including baseline urea, creatinine, electrolytes, urine analysis, complete blood count, coagulation profile, liver functions test, arterial blood gas, serum lactate and daily follow up urea, creatinine, and electrolytes.
4. ECG, echocardiography, and lung ultrasound.
5. Volume status will be assessed by urine output, CVP, mean arterial pressure.
6. The following work up.

   * VExUS score (IVC assessment, hepatic venous, intrarenal venous Doppler and portal vein Doppler)
   * Cardiorenal patient will receive diuretic therapy as a standard treatment in patients with VEXSUS score 1-3
   * Daily VExUS score will be done
   * Diuretic resistance will be defined as failure to produce 0.5 ml/kg/h of urine after administration of at least double the dose of the patient's home diuretic therapy or after administration of 250 mg of Lasix and 10 mg of Metolazone in diuretic naïve patient).

ELIGIBILITY:
Inclusion Criteria:

* Patients with congestive heart failure and GFR less than 100 ml/minute

Exclusion Criteria:

* Patients below 18 years old. Patients with liver cirrhosis and portal hypertension. Patients with IVC thrombus. Patients with inadequate ultrasonography window.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cardiorenal patients above 18 years old
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
response to diuretic | Baseline
  Response to diuretic therapy in cardiorenal patients (failure to produce 0.5 ml/kg/h of urine after administration of at least double the dose of the patient's home diuretic therapy or after administration of 250 mg of Lasix and 10 mg of Metolazone in diuretic naïve patientfailure to produce 0.5 ml/kg/h of urine after administration of at least double the dose of the patient's home diuretic therapy or after administration of 250 mg of Lasix and 10 mg of Metolazone in diuretic naïve patient)

SECONDARY OUTCOMES:
Length of ICU stay | Through study completion, an average of 2 weeks
  Length of ICU stay
Worsening renal function | Through study completion, an average of 2 weeks
  Measurement of Urea and Creatinine on admission and daily follow up Follow up the fluid chart daily (urine input and output) Calculation of eGFR using Cockcroft-Gault Formula on admission daily follow up
Need to ultrafiltration | Baseline
  Patient with symptoms and signs of pulmonary congestion with failure to respond to diuretic therapy and need for ultrafiltration session

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah I. Kelany, MD, Study Director — university

REFERENCES:
- [Background] Rangaswami J, Bhalla V, Blair JEA, Chang TI, Costa S, Lentine KL, Lerma EV, Mezue K, Molitch M, Mullens W, Ronco C, Tang WHW, McCullough PA; American Heart Association Council on the Kidney in Cardiovascular Disease and Council on Clinical Cardiology. Cardiorenal Syndrome: Classification, Pathophysiology, Diagnosis, and Treatment Strategies: A Scientific Statement From the American Heart Association. Circulation. 2019 Apr 16;139(16):e840-e878. doi: 10.1161/CIR.0000000000000664. PMID 30852913
- [Background] Zhang L, Chen Z, Diao Y, Yang Y, Fu P. Associations of fluid overload with mortality and kidney recovery in patients with acute kidney injury: A systematic review and meta-analysis. J Crit Care. 2015 Aug;30(4):860.e7-13. doi: 10.1016/j.jcrc.2015.03.025. Epub 2015 Apr 9. PMID 25979272
- [Background] Rola P, Miralles-Aguiar F, Argaiz E, Beaubien-Souligny W, Haycock K, Karimov T, Dinh VA, Spiegel R. Clinical applications of the venous excess ultrasound (VExUS) score: conceptual review and case series. Ultrasound J. 2021 Jun 19;13(1):32. doi: 10.1186/s13089-021-00232-8. PMID 34146184
- [Background] Bhardwaj V, Vikneswaran G, Rola P, Raju S, Bhat RS, Jayakumar A, Alva A. Combination of Inferior Vena Cava Diameter, Hepatic Venous Flow, and Portal Vein Pulsatility Index: Venous Excess Ultrasound Score (VEXUS Score) in Predicting Acute Kidney Injury in Patients with Cardiorenal Syndrome: A Prospective Cohort Study. Indian J Crit Care Med. 2020 Sep;24(9):783-789. doi: 10.5005/jp-journals-10071-23570. PMID 33132560
- [Background] Shimada S, Hirose T, Takahashi C, Sato E, Kinugasa S, Ohsaki Y, Kisu K, Sato H, Ito S, Mori T. Pathophysiological and molecular mechanisms involved in renal congestion in a novel rat model. Sci Rep. 2018 Nov 14;8(1):16808. doi: 10.1038/s41598-018-35162-4. PMID 30429498
- [Background] Neal CR, Arkill KP, Bell JS, Betteridge KB, Bates DO, Winlove CP, Salmon AHJ, Harper SJ. Novel hemodynamic structures in the human glomerulus. Am J Physiol Renal Physiol. 2018 Nov 1;315(5):F1370-F1384. doi: 10.1152/ajprenal.00566.2017. Epub 2018 Jun 20. PMID 29923763